CLINICAL TRIAL: NCT03481946
Title: A Phase 1 Study to Assess Pharmacokinetics and Pharmacodynamics Following Administration of BAY1093884 in Patients With Severe Hemophilia
Brief Title: A Study to Assess Pharmacokinetics and Pharmacodynamics Following Administration of BAY1093884 in Patients With Severe Hemophilia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19592
Record Dates: First submitted 2018-03-12; First posted 2018-03-29 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BAY1093884 in subjects with Hemophilia (Experimental): Single dose of BAY1093884 over 30 minutes administered in subjects with severe congenital Hemophilia A or B, with inhibitors or without inhibitors
  Interventions: Drug: BAY1093884

INTERVENTIONS:
Drug: BAY1093884 — 0.3 mg/kg given intravenously
Drug: BAY1093884 — 1 mg/kg given intravenously

SUMMARY:
The primary objective of this study is to assess the pharmacokinetics in patients with severe hemophilia.

The secondary objective is to assess the pharmacodynamics of BAY1093884 based on tissue factor pathway inhibitor activity

ELIGIBILITY:
Inclusion Criteria:

* Males with severe congenital hemophilia A or B defined as <1% FVIII or <2% FIX concentration by measurement at the time of screening or from reliable prior documentation (e.g., measurement in other clinical Bayer trials, or diagnostic genetic testing)
* Male with any inhibitor titer at screening or prior to screening at any time from medical records. Subjects may be receiving a bypassing agent (rFVIIa; NovoSeven and/or aPCC; FEIBA) for treatment.
* Age: 18 to 65 years at screening
* BMI: 18 to 29.9 kg/m2

Exclusion Criteria:

* Subjects with known bleeding disorders (such as von Willebrand factor [vWF] deficiency, FXI deficiency, platelet disorders, or known acquired or inherited thrombophilia etc.) other than congenital Hemophilia A or B with or without inhibitors
* History of angina pectoris or treatment for angina pectoris
* History of coronary and/or peripheral atherosclerotic disease, congestive heart failure, disseminated intravascular coagulopathy, or stage 2 hypertension defined as systolic blood pressure (SBP) ≥160 mmHg or diastolic blood pressure (DBP) ≥100 mmHg even if controlled
* History of thrombophlebitis, venous/arterial thromboembolic diseases (particularly deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction, cerebrovascular accident, ischemic heart disease, transient ischemic attack)
* Known or suspected hypersensitivity of the immune system, history of anaphylactic reaction, known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Subjects with inhibitors treated with FEIBA, who are not willing to accept rFVIIa (NovoSeven) for the treatment of any bleeds occurring either between screening and dosing or after study drug administration, and until the end of the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
AUC (0-tlast) of BAY1093884 in plasma | Up to 15 days after drug administration
  Area under the concentration vs. time curve from time 0 to the last data point > LLOQ
AUC(0-tlast)/D of BAY1093884 in plasma | Up to 15 days after drug administration
  AUC(0-tlast) divided by dose
Cmax of BAY1093884 in plasma | Up to 15 days after drug administration
  Maximum observed drug concentration in measured matrix after single dose administration
Cmax/D of BAY1093884 in plasma | Up to 15 days after drug administration
  Cmax divided by dose

SECONDARY OUTCOMES:
Tissue factor plasma inhibitor activity: effect of BAY1093884 to inhibit the anticoagulatory activity of plasma TFPI as assessed by a chromogenic assay | Up to 15 days after drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel